CLINICAL TRIAL: NCT03786874
Title: "Impact of a Programme to Improve Interaction Among Professionals on the Management of Task Interruptions"
Acronym: IMPACTT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC18_0047
Record Dates: First submitted 2018-12-11; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Quality of Life
Keywords: Risk management; health & safety; task interruptions; teamwork

STUDY DESIGN:
Intervention Model Description: Case group:
  Healthcare teams benefiting first the implementation of the coaching model other (centered round the following steps: identify, understand and act) : just after the first measure
  Control group:
  Healthcare teams benefiting first the implementation of the coaching model (centered round the following steps: identify, understand and act) : after the second measure (impact of the device on case group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20 teams the first year (G1) (Active Comparator): control group
  Interventions: Other: Identify work interruptions; Other: Understand work interruptions
- 20 teams second year (G2) (Experimental): case group with implementation of the multi-unit team accompaniment intervention.
  Interventions: Other: Identify work interruptions; Other: Understand work interruptions; Other: Act to limited work interruptions

INTERVENTIONS:
Other: Identify work interruptions — estimate baseline characteristics of the collaborative working model (proportion expressed as a percentage)
Other: Understand work interruptions — Team-review of the results of the task interruption and professional representations, identify activities to protect from task interruption
Other: Act to limited work interruptions — Adaptation of organizations; Awareness raising and Coaching for change
  Arms: 20 teams second year (G2)

SUMMARY:
In 2017, all IMPACTT investigators experimented in coordinated manner on multifacet intervention program, proposed by the present research protocol, with 2 teams from healthcare units from the PDL region. This experiment followed collaborative work aiming to raise team awareness on task interruptions. Given the existing data in the literature, the investigators hypothesise that the implementation of a multifacet program focusing on interactions within a team could enable the percentage of task interruptions linked to interactions between coordination functions and healthcare provision activities to be decreased by 33%. This decrease would concern task interruptions that are avoidable, in order to improve healthcare safety and teamwork.

Also, the main objective of this project is to measure the impact of a program on the evolution of the characteristics of avoidable task interruptions. The project combines quantitative data (observations, questionnaire) and qualitative data (interviews).

DETAILED DESCRIPTION:
This research is a controlled, randomised, blind, pragmatic intervention study (36 months). From the list of volunteering teams meeting inclusion criteria, a random selection will be made. This will enable the formation of two groups of 20 teams each (control group and experimental group). An observational method coupled with a validated questionnaire transfer will allow teams to be questioned about their avoidable task interruptions (control group and experimental group).

The multifacet intervention program is based the concept of teamwork implementation. Targeting potential for improvement will be decided and implemented by each team (experimental group).

Statistics analysis will be conducted on teams before and after the implementation of the program. The assessment criteria will be: the evolution of characteristics of the task interruptions observed (interactions between coordination functions and care delivery functions, prevalence, avoidability, duration, resumption of tasks, social representations of task interruptions).

ELIGIBILITY:
Inclusion Criteria:

* volunteering healthcare teams from healthcare centres in the PDL region,
* public and private legal statuses;
* with at least one activity in standard medical and/or surgical hospitalisation unit,
* agreeing to take part in the project,
* formalising their commitment to the multifacet program (see section 4),
* including 50 professionals at the most,
* including at least the following professional categories: medical, paramedical, administrative, managerial and medical-technical/psycho-social.

Exclusion Criteria:

* Healthcare teams who do not belong to a healthcare unit in the PDL region
* Healthcare teams who do not work in a medical and/or surgical hospitalisation unit.
* Paediatric healthcare teams
* Teams that have already been subjected to a methodological support program from one of the co-investigating units on how to manage task interruptions,
* Teams that do not meet the criteria for commitment to the multifacet program
* Teams of more than 50 members
* Teams who do not include the following professional categories: medical, paramedical, administrative, managerial, medical-technical/psycho-social.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
proportion of avoidable task interruptions | 1 year
  Results from Dual Perspectives Method (DPM)
sources and frequencies of task interruptions | 1 year
  Results from Auto-administered questionnaire (TAA-KH-S)

SECONDARY OUTCOMES:
prevalence of task interruptions | 1 year
  Time measurement of the duration of task interruption upon restart of work

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Teigne D, Cazet L, Mabileau G, Terrien N. Task interruptions from the perspective of work functions: The development of an observational tool applied to inpatient hospital care in France The Team'IT tool. PLoS One. 2023 Mar 9;18(3):e0282721. doi: 10.1371/journal.pone.0282721. eCollection 2023. PMID 36893207